CLINICAL TRIAL: NCT04143438
Title: Assessment of Surgical Correction of Patello-femoral Instability by EOS 3D Kinematics
Acronym: EOS-FP2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL17_0383; UF 9892 (Other: CHU de Montpellier)
Record Dates: First submitted 2019-10-22; First posted 2019-10-29 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2020-06

CONDITIONS: Patellofemoral Dislocation
Keywords: patella; EOS 3D imaging
MeSH Terms: conditions — Patella Fracture | interventions — Postoperative Period

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Undergoing EOS 3D imaging (Experimental): Patients with patello-femoral instability will undergo EOS 3D Imaging protocol before and after undergoing corrective surgery
  Interventions: Procedure: EOS 3D imaging protocol pre- and post-surgery

INTERVENTIONS:
Procedure: EOS 3D imaging protocol pre- and post-surgery — Patients will undergo a EOS 3D Imaging protocol before and 6 months after undergoing patello-femoral surgery. This protocol is already used routinely in the hospital before every patello-femoral surgery.

SUMMARY:
Assessment of surgical correction of patello-femoral instability by EOS 3D kinematics

DETAILED DESCRIPTION:
Patella instability induces repetitive patella dislocation, which impairs day-to-day life. Surgery is commonly used to stabilise the patella during knee flexion. However proofs of efficacy of surgery on patello-femoral kinematics have not yet been found. Analysis of the patello-femoral kinematics is crucial to understand, assess et correct the patella instability. The investigators have developed, validated and published a 3D analysis method from biplanar X-rays (EOS 3D imaging). Our aim in this study is to assess the correction of the patello-femoral kinematics after surgery using the EOS 3D imaging method.

ELIGIBILITY:
Inclusion Criteria:

* Age above 15 years and 3 months (minimal age to be allowed for adult orthopedic surgery in the hospital)
* Patients with patello-femoral instability (at least one patella dislocation)
* Patients with corrective surgery planned
* Patients must be covered by public health insurance
* Signed informed consent form by the patient or by the parents or legal guardian of the patient (if patient is under 18)

Exclusion Criteria:

* Previous existing surgery for patella instability on the same knee
* Previous existing surgery on the extensor apparatus of the knee
* Female patients with pregnancy
* Patients deprived of liberty by administrative or court order

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison of patella lateral tilt before and after surgery | During the presurgery appointment and up to 6 months after surgery
  Efficacy of corrective surgery on patello-femoral instability will be assessed by measuring the patella lateral tilt (Ry) with the knee bending at 0, 20 and 45 degrees, before and after surgery. This measurement will be done using the EOS 3D Imaging technique.

SECONDARY OUTCOMES:
Comparison of patella secondary shifts before and after surgery | During the presurgery appointment and up to 6 months after surgery
  Anterior (Tx), distal (Ty) and lateral (Tz) patella shifts, with the knee bending at 0, 20 and 45 degrees will be measured, before and after surgery. This measurement will be done using the EOS 3D Imaging technique.
Comparison of patella secondary rotations before and after surgery | During the presurgery appointment and up to 6 months after surgery
  External (Rx) and flexion (Rz) rotation of the patella, with the knee bending at 0, 20 and 45 degrees will be measured, before and after surgery. This measurement will be done using the EOS 3D Imaging technique.
Assessment of functional and life quality changes pre- and post-surgery | During the presurgery appointment and up to 6 months after surgery
  The Kujala score and 12-Item Short Form Survey (SF12) life quality questionnaire will be answered by the participants before and after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Louis DAGNEAUX, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dagneaux L, Thoreux P, Eustache B, Canovas F, Skalli W. Sequential 3D analysis of patellofemoral kinematics from biplanar x-rays: In vitro validation protocol. Orthop Traumatol Surg Res. 2015 Nov;101(7):811-8. doi: 10.1016/j.otsr.2015.07.017. Epub 2015 Oct 26. PMID 26514850